CLINICAL TRIAL: NCT06677099
Title: Electrical Impedance Tomography in Guiding Early and Precise Rehabilitation of Patients with Difficult Ventilator Weaning:A Single-cente Randomised Controlled Trial
Brief Title: Electrical Impedance Tomography in Guiding Early and Precise Rehabilitation of Patients with Difficult Ventilator Weaning
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-030
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Difficult-to-Wean Patients
Keywords: mechanical ventilation; electrical impedance tomography

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): Two sessions of CPT (morning and afternoon, 20 minutes each) were conducted. The CPT session consisted of modified postural drainage, assisted cough technique, positive expiratory pressure and chest percussion, vibration. The appointed therapist performed pulmonary auscultation and thoracic palpation to assess the status of pulmonary ventilation and secretion retention, and whether the patient's cough ability can complete effective airway clearance. Individualized program was formed according to the assessment, internal guidelines, the patient's tolerance, education level, and patient's preference prior to the randomization. All CPT sessions were performed by the same physiotherapist to avoid potential bias.
  Interventions: Procedure: chest physiotherapy
- EIT-guided group (Experimental): EIT-guided group: Similar to the patients in the Control group, the CPT techniques were predefined for the patients according to the assessment prior to the randomization. For each CPT session, EIT measurement was conducted and the images were used to guide the CPT treatments. The uses of EIT to guide individual treatments are briefly described as follows.
  Interventions: Procedure: EIT-guided chest physiotherapy

INTERVENTIONS:
Procedure: chest physiotherapy — Two sessions of CPT (morning and afternoon, 20 minutes each) were conducted. The CPT session consisted of modified postural drainage, assisted cough technique , positive expiratory pressure and chest percussion, vibration. The appointed therapist performed pulmonary auscultation and thoracic palpation to assess the status of pulmonary ventilation and secretion retention, and whether the patient's cough ability can complete effective airway clearance. Individualized program was formed according to the assessment, internal guidelines, the patient's tolerance, education level, and patient's preference prior to the randomization. All CPT sessions were performed by the same physiotherapist to avoid potential bias.
  Arms: Control group
Procedure: EIT-guided chest physiotherapy — EIT-guided modified postural drainage combined with vibrations and chest percussion: tidal variation images in EIT reveals heterogeneously ventilated regions. Physiotherapist identified such regions at the bedside and instructed the patient to take the appropriate drainage position, so that the poorly ventilated regions became gravity non-dependent regions. Subsequently, the physiotherapist put her hands on the poorly ventilated area with a vibratory force. A compressive pressure was produced by the therapist's arms.
  Arms: EIT-guided group

SUMMARY:
Diaphragm dysfunction, ineffective chest wall and respiratory muscle function are frequently observed in critically ill patients with difficult weaning from mechanical ventilation(MV).It is the leading cause of retention of airway secretions and insufficient airway clearance.Thechest physiotherapy (CPT) of critically ill patients can reduce secretion retention. We designed a protocol to investigate the feasibility and efficacy of CPT guided by electrical impedance tomography (EIT) in Difficult-to-Wean patients.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation patients who are ≥18 years old, are received to invasive mechanical ventilation more than 96 hours before randomization, are meted the preconditions for the machine to be withdrawn, and at least have one failed attempt to withdraw the ventilator (re-need ventilator support within 48 hours after extubation),
* willing to participate in the study and sign the informed consentsent.

Exclusion Criteria:

* Malignant arrhythmia or acute myocardial ischemia
* Pneumothorax, pulmonary bulla and barotrauma and other lung diseases
* Hemorrhagic disease or abnormal coagulation mechanism with bleeding tendency
* Chest skin trauma
* Pulmonary hypertension and pulmonary embolism
* With a permanent or temporary pacemaker
* There is malignant tumor
* Present and previous history of neuromuscular diseases affecting respiratory muscle
* Participated in another clinical study related to mechanical ventilation withdrawal
* Can not cooperate with the study for any reason or the researcher thinks that it is not suitable to be included in this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
peak expiratory flow | All data will be recorded at the baseline (T1), 14 days (T2) and 28 days (T3)

SECONDARY OUTCOMES:
The cumulative incidence of successful weaning by Day 30 | from admission to discharge, assessed up to 1 day
Maximum inspiratory pressure | All data will be recorded at the baseline (T1), 14 days (T2) and 28 days (T3)
Diaphragm thickening rate | All data will be recorded at the baseline (T1), 14 days (T2) and 28 days (T3)
Diaphragmatic excursion | All data will be recorded at the baseline (T1), 14 days (T2) and 28 days (T3)
Length of ICU stay | from admission to discharge, assessed up to 1 day
Cumulative incidence for death before successful weaning | from admission to discharge, assessed up to 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ge, Principal Investigator — Beijing Rehabilitation Hospital of Capital Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Xi J, Jiang H. Randomized clinical study of electrical impedance tomography-guided chest physiotherapy in difficult-to-wean patients: study protocol. PeerJ. 2025 Aug 4;13:e19727. doi: 10.7717/peerj.19727. eCollection 2025. PMID 40777077